CLINICAL TRIAL: NCT02986113
Title: Men and Providers Preventing Suicide (MAPS): A Randomized Controlled Trial
Brief Title: Men and Providers Preventing Suicide (MAPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 922468; U01CE002664 (NIH)
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Suicidal Intention; Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Men and Providers Preventing Suicide (Experimental): Tailored interactive multimedia intervention, aimed at activating suicidal middle-aged men to disclose and discuss their suicide thoughts with and be receptive to treatment offers from a primary care provider during a linked office visit
  Interventions: Behavioral: MAPS tailored multimedia patient activation program; Behavioral: Telephone evidence-based follow-up care; Behavioral: Commitment to Living for Primary Care
- Sleep hygiene video (Active Comparator): A brief (3 minute) video regarding sleep hygiene, accompanied by introductory text summarizing research linking sleep problems with increased suicide risk.
  Interventions: Behavioral: Sleep hygiene video; Behavioral: Telephone evidence-based follow-up care; Behavioral: Commitment to Living for Primary Care

INTERVENTIONS:
Behavioral: MAPS tailored multimedia patient activation program
  Arms: Men and Providers Preventing Suicide
Behavioral: Sleep hygiene video — 3 minute video on sleep hygiene produced by HealthiNation
  Arms: Sleep hygiene video
Behavioral: Telephone evidence-based follow-up care — 3 months of suicide-focused collaborative mental health care, directed by a supervising psychiatrist and implemented by a care manager working with the patient and their primary care provider
  Other Names: TEBFC
Behavioral: Commitment to Living for Primary Care — Brief (30 minutes total time) video modules presenting participating patients' primary care providers with a patient-centered framework for suicide risk assessment and intervention

SUMMARY:
This study will determine if suicidal middle-aged men who use a personalized computer program addressing suicide risk before a primary care visit are more likely to discuss suicide and accept treatment, reducing their suicide preparatory behaviors and thoughts.This is important because half of all men who die by suicide visit primary care within a month of death, yet few broach the topic, missing chances for prevention.

DETAILED DESCRIPTION:
In this study, the investigators will enroll middle-aged men with active suicide thoughts in a randomized controlled trial (RCT) to examine whether their use of the Men and Providers Preventing Suicide (MAPS) tailored interactive multimedia patient activation program immediately before a primary care provider (PCP) visit, linked with integrated telephone evidence-based follow-up care (TEBFC) (vs. attention control exposure linked with TEBFC), reduces suicide preparatory behaviors and ideation over 3 months. About half of all middle-aged men who die by suicide are seen by a PCP within a month of dying, suggesting the value of primary care-based suicide prevention efforts, to complement strategies in other settings. Current impediments to primary care-based prevention are that many suicidal middle-aged men do not visit a PCP, and among those who do the topic of suicide is rarely broached, due to societal gender-linked norms (e.g., toughness); stigma; spurious concerns that talking about suicide increases risk; competing time demands; and lack of resources to cope with positive responses. PCP-targeted educational interventions have increased detection of suicidal men, but have inconsistently affected suicide behaviors, and still many suicidal men went undetected. Suicide behaviors are more likely to be reduced by evidence-based follow-up care - supportive follow-up contact and collaborative mental health care. However, such care can only be effective if at-risk men visit a PCP who identifies suicide risk and offers the care, and the men accept it. Thus, there is a pressing need to study the use of innovative tools like MAPS to activate at risk middle-aged men to signal their receptiveness to suicide discussion and care, prompting PCP inquiry and referrals to a form of follow-up care that is feasible for most practices to implement (e.g., TEBFC).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified male gender
* Aged 35-74
* Has a PCP at a primary care office in one of the two participating health systems who is actively enrolled in the RCT
* Active suicide thoughts within past 4 weeks
* Able to read and speak English; and self-reported adequate vision, hearing, and hand function to engage with an interactive computer program on a touchscreen electronic tablet device.

Exclusion Criteria:

* Reported or apparent highly unstable medical status (e.g. acute decompensated heart failure requiring immediate care)
* Reported or apparent highly unstable mental health status (e.g. acute uncontrolled psychosis)
* Presence of terminal illness with death anticipated within 3 months
* Plan to leave the current primary care office (e.g., transfer care) within 3 months
* Incarcerated
* Inability to understand and/or provide informed consent, following appropriate explanation

Ages: 35 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2016-12; Primary Completion 2019-07 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Patient: Beck Scale for Suicide Ideation | 3 months

SECONDARY OUTCOMES:
Patient: Reported discussion of suicide during study visits | Immediately post-study visit
Patient: suicidal intent scale | 3 months
Patient: enrollment in telephone evidence-based follow-up care | Immediately post-study visit, 1 month, 2 months, 3 months
Patient adherence to telephone evidence-based follow-up care, ascertained from care manager patient contact logs | 1 month, 2 months, 3 months
Patient: Interpersonal Needs Questionnaire | 1 month, 2 months, 3 months
  Perceived burdensomeness and belongingness to others
Patient: augmented Patient Health Questionnaire (PHQ-9) | 1 month, 2 months, 3 months
  PHQ-9 plus six "male depression" items
Patient: Short Form-12 health survey (SF-12) Mental Component Summary score | 1 month, 2 months, 3 months
  Mental health status
Patient: SF-12 Physical Component Summary score | 1 month, 2 months, 3 months
  Physical health status
Patient: Toughness scale | 1 month, 2 months, 3 months
  Gender-linked views regarding health-related help-seeking
Patient: perceptions of the study interventions and trial participation questionnaire | 3 months
PCP: perceptions of baseline training videos questionnaire | Immediately after completing the video training
  Measured by questionnaire
PCP: reported discussion of suicide during study visits | Immediately post-study visit
PCP: The number of times that PCPs refer study patients to TEBFC, ascertained from study care manager logs | Through study completion, up to 3 years
PCP: attitudes toward caring for suicidal patients questionnaire | At study completion, up to 3 years
PCP: perceptions of study participation questionnaire | At study completion, up to 3 years

OTHER OUTCOMES:
Patient: suicide attempts from electronic medical record and insurance claims database review | Up to 3 years follow-up
The number of times that the trial standardized and proactive safety protocols for patients found to be at heightened acute risk of suicide are invoked, ascertained from patient contact tracking sheets | Through study completion, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Jerant, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - University of California Davis Health System, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jerant A, Duberstein PR, Kravitz RL, Kleiman EM, Rizvi SL, Cipri C, Liu D, Scher L, Freitas M, Jones-Hill M, Oravetz A, Van Orden KA, Franks P. Ethical and methodological challenges slowing progress in primary care-based suicide prevention: Illustrations from a randomized controlled trial and guidance for future research. J Psychiatr Res. 2022 Oct;154:242-251. doi: 10.1016/j.jpsychires.2022.07.038. Epub 2022 Aug 6. PMID 35961180